CLINICAL TRIAL: NCT01339182
Title: A Randomized, Open-label, Single-dose, Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Pegylated-Somatropin in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Pegylated-Somatropin in Healthy Volunteers
Acronym: Somatropin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TB1010GH
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: somatropin; PK; PD; male; pharmacokinetics; pharmacodynamics; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Pegylated-Somatropin, 10mcg/kg (Experimental)
  Interventions: Drug: Pegylated-Somatropin
- Pegylated-Somatropin, 30mcg/kg (Experimental)
  Interventions: Drug: YPEG-Somatropin
- Pegylated-Somatropin, 60mcg/kg (Experimental)
  Interventions: Drug: YPEG-Somatropin
- Pegylated-Somatropin, 120mcg/kg (Experimental)
  Interventions: Drug: YPEG-Somatropin
- Pegylated-Somatropin, 200mcg/kg (Experimental)
  Interventions: Drug: YPEG-Somatropin

INTERVENTIONS:
Drug: Pegylated-Somatropin — Daily s.c, randomized with Saizen, 0.1IU/kg or 0.15IU/kg for the first week, followed by one week wash-out, and then s.c, single dose of pegylated-Somatropin, 10mcg/kg.
  Arms: Pegylated-Somatropin, 10mcg/kg
Drug: YPEG-Somatropin — Daily s.c, randomized with Saizen, 0.1IU/kg or 0.15IU/kg for the first week, followed by one week wash-out, and then s.c, single dose of pegylated-somatropin, 30mcg/kg.
  Arms: Pegylated-Somatropin, 30mcg/kg
Drug: YPEG-Somatropin — Daily s.c, randomized with Saizen, 0.1IU/kg or 0.15IU/kg for the first week, followed by one week wash-out, and then s.c, single dose of pegylated-somatropin, 60mcg/kg.
  Arms: Pegylated-Somatropin, 60mcg/kg
Drug: YPEG-Somatropin — Daily s.c, randomized with Saizen, 0.1IU/kg or 0.15IU/kg for the first week, followed by one week wash-out, and then s.c, single dose of pegylated-somatropin, 120mcg/kg.
  Arms: Pegylated-Somatropin, 120mcg/kg
Drug: YPEG-Somatropin — Daily s.c, randomized with Saizen, 0.1IU/kg or 0.15IU/kg for the first week, followed by one week wash-out, and then s.c, single dose of pegylated-somatropin, 200mcg/kg.
  Arms: Pegylated-Somatropin, 200mcg/kg

SUMMARY:
This study is aimed to assess the safety, tolerability, pharmacokinetics, pharmacodynamics of a single-dose of Pegylated-Somatropin in healthy male volunteers, and collect scientific data for the design and conduct of subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age(yr)between 18 and 45
* Body mass index(BMI)between 20 and 28
* sign informed consent

Exclusion Criteria:

* Known hypersensitivity to somatropin or any other components of the study drug
* Organic lesion in heart, liver, kidney or any other major organs
* History of diabetes mellitus, cancer, autoimmune disease, genetic disease, mental disease
* Alcoholic, smokers or drug abusers
* Blood donation, or massive blood loss due to injury or surgery within 3 months
* Other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the IGF-1 levels for pharmacodynamics study | baseline, one week after initiation of the control drug and two weeks after initiation of the study drug

SECONDARY OUTCOMES:
Measuring the drug levels in blood samples | baseline, one week after initiation of the control drug and two weeks after initiation of the study drug
Measurement of IGFBP-3 levels for pharmacodynamic study | baseline, one week after initiation of the control drug and two weeks after initiation of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Hu Pei, Ph.D, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China